CLINICAL TRIAL: NCT01828723
Title: A Phase One, Open Label, Single Arm Study to Demonstrate the Safety of Antria Cell Preparation Process During Facial Fat Grafting Assisted With Autologous, Adipose Derived Stromal Vascular Fraction (SVF)
Brief Title: Safety Study of Antria Cell Preparation Process to Enhance Facial Fat Grafting With Adipose Derived Stem Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antria (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSVF0001
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Lipoatrophy; Aging; Wrinkles
Keywords: Autologous Adult Stem Cell; Adipose Derived Stem Cell; Stromal Vascular Fraction; SVF; Antria; Shah Rahimian; Leonard Maliver; David Bizousky; Rahul Gore; Lee Quist; Dudley McNitt
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SVF-Enriched Lipoinjection (Experimental)
  Interventions: Biological: SVF

INTERVENTIONS:
Biological: SVF

SUMMARY:
The primary purpose of this study is to demonstrate the safety of injecting the Stromal Vascular Fraction (SVF) [containing Adipose Derived Stem Cells (ADSCs)] enriched fat grafts into regions of the face that require enhancement. The safety of SVF will be evaluated throughout the course of the study phase through the assessment of laboratory values, physical examinations, adverse events, safety phone calls etc.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, Age 18 years or older
2. Subjects that are scheduled for liposuction and facial fat grafting procedures for cosmetic purposes
3. Facial volume defects which could be treated with a total graft volume of between 1mL and 50mL
4. BMI between and including 23 and 28
5. Able to understand and provide written and verbal informed consent

Exclusion Criteria:

1. Currently taking or have taken NSAIDs within last two weeks or corticosteroids within the last six weeks prior to screening
2. Diagnosis of any of the following medical conditions:

   * Active malignancy (diagnosed within 5 years), except for treated non-melanoma skin cancer or other non-invasive or in-situ neoplasm
   * Active infection
   * Type I or Type II Diabetes
3. Subjects who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits, dementia, and/or otherwise considered by the Investigator to be unlikely to complete the study)
4. Subjects with a known drug or alcohol dependence within the past 12 months as judged by the Investigator
5. Subjects with major illnesses involving the renal, hepatic, cardiovascular, and/or nervous systems
6. Subjects with elevated kidney and/or liver functions
7. Any other disease condition or laboratory results that in the opinion of the investigator may be clinically significant and render the subject inappropriate for the study procedure(s), may alter the accuracy of study results, or increase risk for subjects.
8. Subjects with life-expectancies less than 9 months
9. Subjects with known collagenase allergies
10. Subjects with idiopathic or drug-induced coagulopathy
11. Pregnant females
12. On radiotherapy or chemotherapy agents
13. Taking strong CYP450 inhibitors such as protease inhibitors (ritonavir, indinavir, nelfinavir, saquinavir), macrolide antibiotics (clarithromycin, telithromycin), chloramphenicol, azole antibiotics (ketoconazole, itraconazole) and nefazodone.
14. Subjects with a history of keloids or hypertrophic scar formations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the administration of a concentrated SVF-enriched fat graft by monitoring the number and types of adverse events, and via physical examinations, vital signs, 12-lead ECGs, blood draws (CBC/LFT/BMP), and urinalysis. | 6 months

SECONDARY OUTCOMES:
To demonstrate the efficacy of the addition of autologous SVF isolated via Antria Cell Preparation Process by observing graft survival time, volume, and quality of facial re-contouring | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Rahimian, MD, PhD, Principal Investigator — Antria Inc.
Locations (1):
- Delmont Surgery Center, Greensburg, Pennsylvania, United States